CLINICAL TRIAL: NCT05265247
Title: A Randomized, Single Blind, Single Center, Single Dose, Two Period, Two Sequence Crossover Bioequivalence Study of Esomeprazole 20 mg Delayed-Release Capsules (Catalent, Guayama) Compared to the Esomeprazole 20 mg Delayed-Release Capsules ([Nexium 24HR] AstraZeneca Södertälje) in Healthy Adult Subjects Under Fasted Conditions
Brief Title: Bioequivalence Study of Esomeprazole 20 Milligram (mg) Delayed-Release Capsules in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 218246
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product/Reference Product (Experimental): Participants will be randomly assigned to receive Esomeprazole 20 mg delayed-release one capsule once daily as oral administration on day 1 of period 1 and will receive Esomeprazole 20 mg delayed-release one capsule (Nexium 24HR) once daily as oral administration on day 1 of period 2. Participants are instructed to consume the entire amount of ambient temperature water (240 milliliter [mL]) along their investigational product. There will be washout period of 7 days between two treatment periods.
  Interventions: Drug: Esomeprazole 20 mg Delayed-Release Capsules; Drug: Esomeprazole 20 mg Delayed-Release Capsules (Nexium 24HR)
- Reference Product/Test Products (Experimental): Participants will be randomly assigned to receive Esomeprazole 20 mg delayed-release one capsule (Nexium 24HR) once daily as oral administration on day 1 of period 1 and will receive Esomeprazole 20 mg delayed-release one capsule once daily as oral administration on day 1 of period 2. Participants are instructed to consume the entire amount of ambient temperature water (240 milliliter [mL]) along their investigational product. There will be washout period of 7 days between two treatment periods.
  Interventions: Drug: Esomeprazole 20 mg Delayed-Release Capsules; Drug: Esomeprazole 20 mg Delayed-Release Capsules (Nexium 24HR)

INTERVENTIONS:
Drug: Esomeprazole 20 mg Delayed-Release Capsules — Esomeprazole 20 mg delayed-release capsules will be given as one capsule once daily as oral administration.
Drug: Esomeprazole 20 mg Delayed-Release Capsules (Nexium 24HR) — Esomeprazole 20 mg delayed-release capsules (Nexium 24HR) will be given as one capsule once daily as oral administration.

SUMMARY:
The purpose of this study is to evaluate bioequivalence parameters of esomeprazole capsules 20 mg (test product) vs. esomeprazole capsules 20 mg (reference product) under fasted conditions.

DETAILED DESCRIPTION:
This will be a single center, single dose, single-blind, randomized, two-sequence, two-period crossover, bioequivalence study in healthy adult participants with at least a 7-day washout period. The study will consist of an ambulant screening day within 28 days prior to first product administration and two study periods.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Healthy Participant, which is defined as in general good physical health, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG) or clinical laboratory tests.
* Body Mass Index (BMI) of 18.5 to 30.0 Kilogram per square meter (kg/m^2); and a total body weight Greater than or equal to (>=) 50.0 kg for males and >=45.0 kg for females.
* Participant with two negative tests (one at screening within 72 hours of admission and one at check on Day-1) for active COVID-19, separated by Greater Than (>) 24 hours.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. Female participants who are not of childbearing potential must meet requirements in the Contraception section of protocol.

Exclusion Criteria:

* Participant who is an investigational site staff member directly involved in the conduct of the study and his/her family members, site staff member otherwise supervised by the investigator, or participant who is a GSK employee directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participant.
* Breastfeeding female participant.
* Known or suspected intolerance or hypersensitivity or photosensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Diagnosis of long QT syndrome or QTc > 450 Millisecond (msec) for males and > 470 msec for females.
* Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 Millimeter of mercury (mmHg), diastolic blood pressure lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 beats per minute (bpm).
* A participant unwilling or unable to comply with Lifestyle Considerations described in this protocol.
* Use of any medication (including over-the-counter medications and herbal remedies) within 2 weeks before first scheduled study drug administration or within less than 10 times the elimination half-life of the respective drug (whichever is longer), or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  * systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study;
  * occasional use of acetaminophen (up to 2 g daily).
* Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* Participant with signs and symptoms suggestive of COVID-19 (i.e. fever, cough, etc)* within 14 days of inpatient admission. *as defined by WHO or local guidance)
* Participant with known COVID-19 positive contacts in the past 14 days.
* Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:

  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, e.g., appendectomy and herniorrhaphy);
  * History of inflammatory bowel disease;
  * History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (> 123 micromole per liter [μmol/L] for males and > 95 μmol/L for females) or blood urea nitrogen (BUN) (>= 12.0 millimoles per liter [mmol/L]) or the presence of clinically significant abnormal urinary constituents (e.g. albuminuria);
  * History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found: 1) aspartate transaminase (AST) (>= 1.2 upper limit of normal [ULN]), alanine transaminase [ALT] (>= 1.2 ULN), 2) gamma-glutamyl transpeptidase (GGT) (>= 1.2 ULN), alkaline phosphatase (ALP) (>= 1.2 ULN), 3) bilirubin (>= 48 μmol/L for males and >= 30 μmol/L for females) or creatine kinase (CK) (>= 3 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the investigator;
  * Evidence of urinary obstruction or difficulty in voiding at screening;
  * History or clinical evidence at screening of pancreatic injury or pancreatitis.
* Participant has a history of drug abuse or investigator has evidence of current drug abuse with drug classes that include but are not limited to barbiturates, tricyclic antidepressants, amphetamines, benzodiazepines, cocaine, opiates, cannabis or any other drugs (verified by urine drug screen or other reliable evidence).
* Evidence, as reported by an alcohol breath testing, for current alcohol abuse or reports a regular average alcohol consumption exceeding 18 g (women) or 35 g (men) of pure alcohol per day, i.e. 1 drink/day for women or 2 drinks/day for men (1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor) within 6 months of screening.
* Participant reported regular consumption of > 5 cups of coffee or tea per day (or equivalent consumption of >= 500 mg xanthine per day using other products)
* Smoker, defined as the use of tobacco or nicotine products during the 3 months prior to screening until admission to the unit or a positive urine cotinine test at screening.
* A participant who is unwilling to abstain from tobacco or nicotine-containing product use during the study.
* Participant reports consumption of any drug metabolizing enzyme (e.g. cytochrome P450 [CYP]3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (e.g. broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort etc.) within 2 weeks prior to screening until admission to the unit.
* Positive results in any of the virology tests for human immunodeficiency virus (HIV) antigen and antibody, hepatitis C virus antibody (HCV Ab), hepatitis B surface antigen (HbsAg), and hepatitis B core antibody (HBcAb) ([immunoglobulin G] IgG + immunoglobulin M [IgM]).
* Performance of unaccustomed strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission and throughout the entire study.
* Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the investigator's opinion may pose a risk to the candidate.
* Any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the participant at risk
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 milliliter (mL) to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dose.
* Participant who has previously been enrolled in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos health, Québec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Canada.
Pre-assignment Details: A total of 61 participants were enrolled, of which 55 participants were randomized and dosed (6 enrolled participants were not randomized).
Groups:
- Esomeprazole CG (Test)/Esomeprazole AZ (Reference): Participants received Esomeprazole 20 milligram (mg) delayed-release from Catalent, Guayama (CG) (Test product) one capsule once daily as an oral administration on day 1 of period 1. Participants received Esomeprazole 20 mg delayed-release (Nexium 24 hour [HR]) from AstraZeneca (AZ) (Reference product) one capsule once daily as an oral administration on day 1 of period 2. Participants received the investigational products in the fasted state with approximately 240 milliliters (mL) of entire amount of ambient temperature water. There was a washout period of at least 7 days between each dosing.
- Esomeprazole AZ (Reference)/Esomeprazole CG (Test): Participants received Esomeprazole 20 mg delayed-release (Nexium 24 hour [HR]) from AZ (Reference Product) one capsule once daily as an oral administration on day 1 of period 1. Participants received Esomeprazole 20 mg delayed-release from CG (Test product) one capsule once daily as an oral administration on day 1 of period 2. Participants received the investigational products in the fasted state with approximately 240 mL of entire amount of ambient temperature water. There was a washout period of at least 7 days between each dosing.
Period: Period 1 (2 Days)
Arm/Group | Esomeprazole CG (Test)/Esomeprazole AZ (Reference) | Esomeprazole AZ (Reference)/Esomeprazole CG (Test)
Started | 26 | 29
Completed | 26 | 29
Not Completed | 0 | 0
Period: Washout Period (7 Days)
Arm/Group | Esomeprazole CG (Test)/Esomeprazole AZ (Reference) | Esomeprazole AZ (Reference)/Esomeprazole CG (Test)
Started | 26 | 29
Completed | 22 | 22
Not Completed | 4 | 7
Not completed — Positive Result for Coronavirus (COVID)-19 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-compliance with study requirements | 3 | 3
Period: Period 2 (2 Days)
Arm/Group | Esomeprazole CG (Test)/Esomeprazole AZ (Reference) | Esomeprazole AZ (Reference)/Esomeprazole CG (Test)
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population- comprised all randomized participants who received at least one dose of study medication.
Groups:
- Esomeprazole CG (Test)/Esomeprazole AZ (Reference): Participants received Esomeprazole 20 mg delayed-release from CG (Test product) one capsule once daily as an oral administration on day 1 of period 1. Participants received Esomeprazole 20 mg delayed-release (Nexium 24 [HR]) from AZ (Reference product) one capsule once daily as an oral administration on day 1 of period 2. Participants received the investigational products in the fasted state with approximately 240 mL of entire amount of ambient temperature water. There was a washout period of at least 7 days between each dosing.
- Esomeprazole AZ (Reference)/Esomeprazole CG (Test): Participants received Esomeprazole 20 mg delayed-release (Nexium 24 [HR]) from AZ (Reference Product) one capsule once daily as an oral administration on day 1 of period 1. Participants received Esomeprazole 20 mg delayed-release from CG (Test product) one capsule once daily as an oral administration on day 1 of period 2. Participants received the investigational products in the fasted state with approximately 240 mL of entire amount of ambient temperature water. There was a washout period of at least 7 days between each dosing.
- Total: Total of all reporting groups
Arm/Group | Esomeprazole CG (Test)/Esomeprazole AZ (Reference) | Esomeprazole AZ (Reference)/Esomeprazole CG (Test) | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (9.63) | 37.0 (10.90) | 38.1 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 25 | 29 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Post Dose Concentration (Cmax)
Description: Cmax is defined as maximum observed post-dose concentration; obtained without interpolation. Blood samples were collected at the indicated time points for the analysis of Cmax. Pharmacokinetic (PK) parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose (within 1 hour prior to dosing), 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8,10, 12, 16, and 24 hours post dose in each treatment period (each period is of 2 days)
Population: PK analysis set included all participants of the PK population who completed both treatment periods, and for which the relevant PK parameters (at least at least Area Under the Plasma Concentration Versus Time Curve Calculated from Time 0 to the Last Measurable Sampling Time Point [AUC0-t] or Cmax) could be derived. Participants with baseline concentration greater than (>) 5 percent (%) of the individual Cmax for either period were to be excluded from the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Groups:
- Esomeprazole CG (Test): Participants received Esomeprazole 20 mg delayed-release from CG (Test product) one capsule once daily as an oral administration on day 1 of period 1 or period 2 as per randomization schedule. Participants received the investigational product in the fasted state with approximately 240 mL of entire amount of ambient temperature water.
- Esomeprazole AZ (Reference): Participants received Esomeprazole 20 mg delayed-release (Nexium 24 [HR]) from AZ (Reference Product) one capsule once daily as an oral administration on day 1 of period 1 or period 2 as per randomization schedule. Participants received the investigational product in the fasted state with approximately 240 mL of entire amount of ambient temperature water.
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 44 | 44
Nanograms per milliliter | 483 (51.1) | 514 (46.2)
Statistical Analysis 1: Comparison: Esomeprazole CG (Test) vs Esomeprazole AZ (Reference); Test type: Equivalence — The two formulations were considered to be bioequivalent if the point estimate for the ratio lies completely within the range of 0.8-1.25; Ratio of Geometric least squares mean = 0.9531, 90% CI 2-sided [0.8510 to 1.0673]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to the Last Measurable Sampling Time Point
Description: AUC(0-t) is defined as area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point t, computed using the linear trapezoidal rule. Blood samples were collected at the indicated time points for the analysis of AUC0-t. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 44 | 44
Hour*nanograms per milliliter | 772.10 (74.0) | 815.55 (68.6)
Statistical Analysis 1: Comparison: Esomeprazole CG (Test) vs Esomeprazole AZ (Reference); Test type: Equivalence — The two formulations were considered to be bioequivalent if the 90% 2-sided confidence interval (CI) for the ratio lies completely within the range of 0.8-1.25; Ratio of Geometric least squares mean = 0.9538, 90% CI 2-sided [0.8980 to 1.0132]

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to Infinity (AUC0-inf)
Description: AUC(0-inf) is defined as area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC0-inf is equal to (=) AUC0-t plus (+) concentration at the last measurable sampling time point [C(t)]/terminal elimination rate constant (λz). Blood samples were collected at the indicated time points for the analysis of AUC0-inf. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants having adjusted coefficient of determination greater than equal to 0.80 for the derived parameter AUC0-inf were included for summary statistics and statistical modelling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 42 | 43
Hour*nanograms per milliliter | 792.72 (73.5) | 800.94 (68.8)

4. Secondary Outcome: Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex)
Description: %AUCex is defined as percentage of AUC(0-inf) obtained by extrapolation, calculated as (1-[AUC{0-t}/AUC{0-inf}]) ×100. Blood samples were collected at the indicated time points for the analysis of %AUCex. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants having adjusted coefficient of determination greater than equal to 0.80 for the derived parameter %AUCex were included for summary statistics and statistical modelling.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC Extrapolated
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 42 | 43
Percentage of AUC Extrapolated | 0.34 (109.1) | 0.35 (74.6)

5. Secondary Outcome: Terminal Elimination Rate Constant
Description: λz is defined as terminal elimination rate constant computed as the slope of the regression line of ln (C[t]) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples were collected at the indicated time points for the analysis of λz. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants having adjusted coefficient of determination greater than equal to 0.80 for the derived parameter λz were included for summary statistics and statistical modelling.
Measure: Median (Full Range); unit: 1 per hour
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 42 | 43
1 per hour | 0.8839 [0.3528 to 1.4328] | 0.8504 [0.3524 to 1.5184]

6. Secondary Outcome: Time of the Maximum Observed Post-Dose Concentration (Tmax)
Description: Tmax is defined as the time of the maximum observed post-dose concentration. Blood samples were collected at the indicated time points for the analysis of Tmax. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: Hour
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 44 | 44
Hour | 1.983 [0.733 to 5.983] | 1.983 [0.983 to 4.483]

7. Secondary Outcome: Elimination Half-Life (T1/2)
Description: T1/2 is defined as elimination half-life computed as T1/2 = ln(2)/ λz. Blood samples were collected at the indicated time points for the analysis of T1/2. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 1
Population: PK analysis set. Only those participants having adjusted coefficient of determination greater than equal to 0.80 for the derived parameter T1/2 were included for summary statistics and statistical modelling.
Measure: Median (Full Range); unit: Hour
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
Number analyzed (Participants) | 42 | 43
Hour | 0.78 [0.48 to 1.96] | 0.82 [0.46 to 1.97]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the signing of informed consent until 5 days after last administration of study product (up to 41 days).
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) is a particular category of an adverse event where the adverse outcome is serious. AEs were presented treatment wise.
Arm/Group | Esomeprazole CG (Test) | Esomeprazole AZ (Reference)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 8/48 | 13/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole CG (Test) (N=48) | Esomeprazole AZ (Reference) (N=51)
Covid-19 (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Red blood cells urine (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT05265247/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05265247/SAP_001.pdf